CLINICAL TRIAL: NCT07234773
Title: A Phase 1a, Open-Label, First-in-Human Study to Investigate the Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of KT501 by a Single Subcutaneous Administration in Participants With Rheumatoid Arthritis
Brief Title: A First-in-human Study of KT501 Administered Subcutaneously to Patients With Rheumatoid Arthritis (RA).
Status: Not yet recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Kali Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: KT501-001
Record Dates: First submitted 2025-11-13; First posted 2025-11-18 (Actual); Last update posted 2025-11-18 (Actual); Status verified 2025-11

CONDITIONS: Rheumatoid Arthritis (RA)
Keywords: Rheumatoid Arthritis (RA); Autoimmune; T-cell Engagers (TCEs); B-cell Depletion
MeSH Terms: conditions — Arthritis, Rheumatoid

STUDY DESIGN:
Intervention Model Description: Single Ascending Dose (SAD)
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | Unapproved Device: Yes | US Export: No

ARMS (5):
- Dose Level 1 (Experimental): KT501 Subcutaneous Injection Dose Level 1
  Interventions: Drug: KT501
- Dose Level 2 (Experimental): KT501 Subcutaneous Injection Dose Level 2
  Interventions: Drug: KT501
- Dose Level 3 (Experimental): KT501 Subcutaneous Injection Dose Level 3
  Interventions: Drug: KT501
- Dose Level 4 (Experimental): KT501 Subcutaneous Injection Dose Level 4
  Interventions: Drug: KT501
- Dose Level 5 (Experimental): KT501 Subcutaneous Injection Dose Level 5
  Interventions: Drug: KT501

INTERVENTIONS:
Drug: KT501 — KT501 is a monoclonal antibody that depletes B cells including plasma cells by targeting CD19, BCMA and CD3.

SUMMARY:
This is a Phase 1, open-label, first-in-human study to investigate the safety, tolerability, pharmacokinetics and pharmacodynamics of KT501 administered subcutaneously to participants with Rheumatoid Arthritis (RA).

DETAILED DESCRIPTION:
This is a Phase 1, open-label, first-in-human dose escalation study to investigate the safety, tolerability, pharmacokinetic and pharmacodynamic of KT501 by a single subcutaneous administration in participants with Rheumatoid Arthritis (RA).

Up to a total of 5 cohorts with up to approximately 14 participants in total with RA will be enrolled. All will receive a single dose of KT501 on Day 1 and followed up until Week 12. For any participants with B cells lower than baseline level or lower limit quantification, whichever is lower, additional B cell follow up is required up to 6 months after the study treatment.

ELIGIBILITY:
Inclusion Criteria:

1. 18 to 75 years old
2. Diagnosis of adult-onset RA for at least 6 months
3. Moderately to severely active RA
4. Inadequate treatment response as defined in the protocol
5. RF + or ACPA+
6. Stable use of traditional DMARDs is permitted
7. Willing and able to comply with all study assessments and adhere to the protocol schedule and restrictions.

Exclusion Criteria:

1. Functional class IV as defined by the ACR Classification of Functional Status in RA
2. Presence of any concomitant autoimmune disease other than RA
3. Active infection, history of serious recurrent or chronic infection
4. History of progressive multifocal leukoencephalopathy
5. Have a diagnosis or history of malignant disease within 5 years or breast cancer diagnosed within the previous 10 years.
6. History of or planned organ transplant and/or autologous or allogeneic hematopoietic stem cell transplantation
7. Receipt of live vaccine within 4 weeks
8. Major surgery (including joint surgery) within 8 weeks prior to screening or planned major surgery within 6 months after study
9. Women who are pregnant or breastfeeding
10. Significant or uncontrolled medical disease that would preclude participant participation

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Estimated)
Dates: Start 2025-12-15 (Estimated); Primary Completion 2027-02 (Estimated); Study Completion 2027-08 (Estimated)

PRIMARY OUTCOMES:
Incidence of Adverse Events | From Baseline Up to 12 weeks
  Incidence and severity of Adverse Events, with severity determined according to National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) v5.0.
Incidence of Cytokine-release Syndrome (CRS) | From Baseline Up to 12 Weeks
  Incidence and severity of CRS with severity determined according to the 2019 American Society for Transplantation and Cellular Therapy (ASTCT) CRS Consensus grading criteria
Changes in Pulse Rate from Baseline | From Baseline Up to 12 Weeks
  Vital signs: Changes in Pulse Rate from Baseline
Changes in Respiratory Rate from Baseline | From Baseline to 12 Weeks
  Vital Signs: Changes in Respiratory Rate from Baseline
Changes in Blood Pressure from Baseline | From Baseline Up to Week 12
  Vital Signs: Changes in Blood Pressure from Baseline
Changes in Temperature from Baseline | From Baseline to 12 Weeks
  Vital Signs: Changes in Body Temperature from Baseline
Changes in Hematology Clinical Laboratory Results from Baseline | From Baseline Up to 12 Weeks
  Hematology: Changes in results from Baseline
Changes in Chemistry Clinical Laboratory Results from Baseline | From Baseline Up to 12 Weeks
  Chemistry: Changes in results from Baseline
Changes in Urinalysis Clinical Laboratory Results from Baseline | From Baseline Up to 12 Weeks
  Urinalysis: Changes in results from Baseline
Changes in Coagulation Clinical Laboratory Results from Baseline | From Baseline Up to 12 Weeks
  Coagulation: Changes in results from Baseline

SECONDARY OUTCOMES:
Serum Concentrations of KT501 | Pre-dose and 6 hours post-dose on Day 1; Day 2, 3, 4, 5, 8, 11, 15, 22, 29, 43, 57 and 85.
  Blood samples will be collected at specific time points for calculating serum concentrations of KT501
Incidence of Treatment-induced Anti-Drug Antibodies (ADAs) | Pre-dose and on Day 1; Day 8, 11, 15, 22, 29, 43, 57 and 85.
  For Immunogenicity: Incidence of participants with treatment induced Anti-Drug Antibodies (ADA)
To Determine Cmax | Day 1 - Day 85
  Maximum observed serum KT501 concentration
To Determine Tmax, Derived from Serum Concentration of each Dose of KT501 | Day 1 - Day 85
  Time to maximum observed concentration
Area Under the Serum-concentration Time Curve (AUC) from Time Zero to the Last Timepoint with Measurable Analyte Concentration (AUC0-t) | Day 1 - Day 85
  Area under the concentration-time curve from 0 to the time of the last quantifiable concentration (AUClast)
AUC from Time Zero to Infinity (AUCinf) | Day 1 - Day 85
  Area under the plasma concentration versus time curve (AUC) from time 0 extrapolated to infinity
To Determine Terminal Half-Life (T1/2) | Day 1 - Day 85
  Terminal elimination half life summarized by dosing regimen
Total Body Clearance (CL/F) | Day 1 - Day 85
  CL is the measure of the rate at which a drug is metabolized or eliminated by normal biological processes
Volume of Distribution During the Terminal Phase (Vz/F) | Day 1 - Day 85
  Vz is defined as the theoretical volume in which the total amount of drug would need to be uniformly distributed to produce the desired serum concentration of a drug.
Change in Levels of B Cell Count | Pre-dose on Day 1; Day 2, 3, 4, 5, 8, 11, 15, 22, 29, 43, 57 and 85.
  Pharmacodynamics: Change in levels of B cell counts measured at specific timepoints
Duration of B Cell Depletion | Day 1 - Day 85
  Pharmacodynamics: The duration of B cell depletion measured from Baseline
Change in Levels of Acute Inflammatory Markers | Pre-dose and 6 hours post-dose on Day 1; Day 2, 3, 4, 5, 8, 15, 22, 29,, 57 and 85.
  Pharmacodynamics: Change in levels of acute Inflammatory markers (C-reactive protein (CRP) and CRS-related cytokines at specific timepoints
Changes in Blood Pressure from Baseline | From Baseline to 12 Weeks
  Vital Signs: Changes in Blood Pressure from Baseline

IPD SHARING:
Plan to Share IPD: No
This is a Phase 1 trial.